CLINICAL TRIAL: NCT05183152
Title: Non-invasive Brain-computer Interfaces for Control of Assistive Devices
Brief Title: Non-invasive BCI-controlled Assistive Devices
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Jose del R. Millan, Professor, University of Texas at Austin
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 2020030073
Record Dates: First submitted 2021-12-20; First posted 2022-01-10 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Motor Disorders; Healthy; Spinal Cord Injuries; Muscular Diseases; Motor Neuron Disease; Stroke; Traumatic Brain Injury; Movement Disorders; Multiple Sclerosis
Keywords: motor deficits; able-bodied, healthy; unilateral and bilateral stroke; spinal cord injury; motor neuron diseases; muscular diseases (i.e. myopathy); traumatic or neurological pain; movement disorders
MeSH Terms: conditions — Motor Disorders; Spinal Cord Injuries; Muscular Diseases; Motor Neuron Disease; Stroke; Brain Injuries, Traumatic; Movement Disorders; Multiple Sclerosis; Neurologic Manifestations

STUDY DESIGN:
Intervention Model Description: BCI Task x Stimulation Modality
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- TESS BCI - Standard MI Task (Experimental): Transcutaneous Electrical Spinal Stimulation (TESS) is applied for 20 minutes prior to BCI training sessions. Following TESS, BCI training is performed with visual feedback contingent to motor imagery as detected by a closed-loop BCI.
  Interventions: Device: Visual Feedback; Device: TESS
- Visual BCI - Standard MI Task (Active Comparator): Conventional BCI training is performed with visual feedback contingent to the imagination of right versus left hand movements as detected by a closed-loop BCI.
  Interventions: Device: Visual Feedback
- NMES BCI - Difficult MI Task (Experimental): BCI training is performed with NMES instead of Visual feedback. NMES is delivered over the flexors/extensors of the forearm contingent to the imagination of same-hand wrist and fingers flexion versus extension as detected by a closed-loop BCI.
  Interventions: Device: NMES Feedback
- Visual BCI - Difficult MI Task (Active Comparator): Conventional BCI training is performed with visual feedback contingent to the imagination of same-hand wrist and fingers flexion versus extension as detected by a closed-loop BCI.
  Interventions: Device: Visual Feedback

INTERVENTIONS:
Device: NMES Feedback — Electroencephalography (EEG) signals will be recorded from subjects as they perform cued tasks for flexing/extending their non-dominant hand. The signals will be processed and classified in real-time using machine learning algorithms to trigger electrical stimulation on the flexors/extensors of the targeted arm contingent to the detection of a subject-specific flexion/extension EEG patterns.
  Arms: NMES BCI - Difficult MI Task
Device: Visual Feedback — Electroencephalography (EEG) - recorded from subjects as they perform cued motor imagery (MI) tasks - are classified in real-time using a subject-specific BCI decoder,. The output classification probability of the decoder is accumulated using exponential smoothing and translated into continuous visual feedback by means of a bar - on a computer screen - that moves to the right or left in response to classification of one or the other MI task.
  Arms: TESS BCI - Standard MI Task; Visual BCI - Difficult MI Task; Visual BCI - Standard MI Task
Device: TESS — Transcutaneous Electrical Spinal Stimulation (TESS) is applied over the C5-C6 spinal segment for 20 minutes at 30Hz with 5kHz carrier frequency.
  Arms: TESS BCI - Standard MI Task

SUMMARY:
Injuries affecting the central nervous system may disrupt the cortical pathways to muscles causing loss of motor control. Nevertheless, the brain still exhibits sensorimotor rhythms (SMRs) during movement intents or motor imagery (MI), which is the mental rehearsal of the kinesthetics of a movement without actually performing it. Brain-computer interfaces (BCIs) can decode SMRs to control assistive devices and promote functional recovery. Despite rapid advancements in non-invasive BCI systems based on EEG, two persistent challenges remain: First, the instability of SMR patterns due to the non-stationarity of neural signals, which may significantly degrade BCI performance over days and hamper the effectiveness of BCI-based rehabilitation. Second, differentiating MI patterns corresponding to fine hand movements of the same limb is still difficult due to the low spatial resolution of EEG. To address the first challenge, subjects usually learn to elicit reliable SMR and improve BCI control through longitudinal training, so a fundamental question is how to accelerate subject training building upon the SMR neurophysiology. In this study, the investigators hypothesize that conditioning the brain with transcutaneous electrical spinal stimulation, which reportedly induces cortical inhibition, would constrain the neural dynamics and promote focal and strong SMR modulations in subsequent MI-based BCI training sessions - leading to accelerated BCI training. To address the second challenge, the investigators hypothesize that neuromuscular electrical stimulation (NMES) applied contingent to the voluntary activation of the primary motor cortex through MI can help differentiate patterns of activity associated with different hand movements of the same limb by consistently recruiting the separate neural pathways associated with each of the movements within a closed-loop BCI setup. The investigators study the neuroplastic changes associated with training with the two stimulation modalities.

ELIGIBILITY:
Inclusion Criteria:

1. Able-bodied participants:

   * good general health
   * normal or corrected vision
   * no history of neurological/psychiatric disease
   * ability to read and understand English (Research Personnel do not speak Spanish)
2. Subjects with motor disabilities

   * motor deficits due to: unilateral and bilateral stroke / spinal cord injury / motor neuron diseases (i.e. amyotrophic lateral sclerosis, spino-cerebellar ataxia, multiple sclerosis) / muscular diseases (i.e. myopathy) / traumatic or neurological pain / movement disorders (i.e. cerebral palsy) / orthopedic / traumatic brain injury / brain tumors
   * normal or corrected vision
   * ability to read and understand English
   * ability to provide informed consent

Exclusion Criteria:

1. Subjects with motor disabilities

   * short attentional spans or cognitive deficits that prevent the subject from concentrating during the whole experimental session
   * heavy medication affecting the central nervous system (including vigilance)
   * concomitant serious illness (e.g., metabolic disorders)
2. All participants

   * factors hindering EEG/EMG acquisition and the delivery of non-invasive electrical stimulation (e.g., skin infection, wounds, dermatitis, metal implants under electrodes)
   * criteria identified in safety guidelines for MRI and TMS, in particular metallic implants

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-16 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in the BCI command delivery performance | immediately after each intervention session and up to one week after all sessions
  The command delivery accuracy reflects the level of control of the subject when using the BCI. It measures the percentage of trials in which the subject-specific classifier that is used to differentiate the different imagined movements could accumulate enough evidence to support the presence of EEG patterns specifically associated with the imagined movement in those trials.
  The score is 0-100, and the higher the value, the better the outcome.
Change in the focality and Strength of SMR Modulation | immediately after each intervention session and up to one week after all sessions
  The focality of sensorimotor rhythm modulation is assessed from EEG using event-related desynchorinzation (ERD) and synchronization (ERS) over the motor area.
  Continuous measure, the higher the better

SECONDARY OUTCOMES:
Stability of Motor Imagery features | immediately after each intervention session and one-day after all sessions
  The features corresponding to different motor imagery tasks become more stable at the end of the intervention.
Separability of Motor Imagery features | immediately after each intervention session and one-day after all sessions
  The features corresponding to different motor imagery tasks become more separable after the intervention.
Changes in motor-evoked potential amplitude | immediately after each intervention session and one-day after all sessions
  Continuous measure, the higher the better
Changes in electroencephalography functional connectivity | immediately after each intervention session and one-day after all sessions
  Continuous measure, the more significant changes the better
Change in focality of fMRI activation for different imagined movements | immediately after each intervention session and one-day after all sessions
  The clusters of significant activation during MI of different movements would be more focal in the associated region of the motor area Continuous measure, the more the better.
More discriminable fMRI activations for different imagined movements | immediately after each intervention session and one-day after all sessions
  The activation associated with different MI tasks would be more discriminable from BOLD signals.
  Continuous measure, the more the better.

CONTACTS AND LOCATIONS:
Overall Officials: Jose del R. Millan, PhD, Principal Investigator — The University of Texas at Austin
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: All data will be made available by the online publication date
Access Criteria: Data will be placed in public servers for any interested researcher to access it